CLINICAL TRIAL: NCT00223769
Title: The Use of Oxandrolone to Improve Function in Persons With Chronic Spinal Cord Injury
Brief Title: The Use of Anabolic Steroids to Improve Function After Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: B2656C
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2008-02-13 (Estimated); Status verified 2006-05

CONDITIONS: Spinal Cord Injury
Keywords: oxandrolone; oxandrin; lean body mass; functional recovery; resistance training
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Oxandrolone

INTERVENTIONS:
Drug: Oxandrolone

SUMMARY:
The purpose of this study is to determine the effect of oxandrolone on the function and quality of life of patients with chronic spinal cord injury.

DETAILED DESCRIPTION:
Spinal cord injury results in significant loss of muscle mass. Oxandrolone, a derivative of testosterone, is an anabolic steroid shown to promote gain in body weight and muscle mass after trauma, severe illness, surgery, burns, and stress. To date there are no studies that have evaluated the effect of oxandrolone in persons with chronic spinal cord injury. This study will assess the effect of oxandrolone on strength, metabolic rate, lean body mass, pulmonary function, and ambulation in persons with chronic SCI. This study has the potential to yield valuable information concerning the use of oxandrolone after SCI.

ELIGIBILITY:
Inclusion Criteria:

Part-A

* Diagnosed with a traumatic injury to spinal cord
* Motor complete injury at level of C5 to T12
* Date of injury at least one year prior to enrollment
* Sufficient upper body strength to participate in a 12-week resistance training program with accommodation for disability in hand strength and/or grasping
* Lean body mass in lower extremities less than 90% of normal as determined by DEXA scan
* Willingness to take study medication for 12 weeks twice a day by mouth

Part-B:

* Diagnosed with a traumatic injury to the spinal cord
* Motor incomplete injury at any level
* Date of injury at least one year prior to enrollment
* Lean body mass in lower extremities less than 90% of normal as determined by DEXA scan
* Ability to stand independently with or without the aid of assistive device(s)
* Willingness to take study medication for 12 weeks twice a day by mouth

Exclusion Criteria:

Active medical problems including:

* Uncontrolled diabetes
* Cardiovascular disease
* Cancer
* Liver disease
* Hypocalcaemia
* Nephritic syndrome
* HIV/AIDS
* Pressure ulcers of grade 3 or 4
* Shoulder pathology
* Pregnancy

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-01; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Part-A: lean body mass, upper extremity muscle strength. Measures are made at baseline, 12-weeks (end of intervention), and at 24-weeks.
Part-B: respiratory function, efficency of ambulaton (speed and quality of gait). Measures are made at baseline,
12-weeks (end of intervention), and at 24-weeks.

SECONDARY OUTCOMES:
Part-A: maximum VO2/respiratory function, functional status, safety, quality of life, community
re-integration.
Part-B: upper extremity strength, lean body mass, functional status, safety, quality of life, community

CONTACTS AND LOCATIONS:
Overall Officials: Kresimir Banovac, PhD MD, Principal Investigator — VA Spinal Cord Injury Service
Locations (1):
- Miami Veterans Affairs Medical Center, Miami, Florida, United States

REFERENCES:
- [Background] Barton RG. Nutrition support in critical illness. Nutr Clin Pract. 1994 Aug;9(4):127-39. doi: 10.1177/0115426594009004127. PMID 8078451
- [Background] Kearns PJ, Thompson JD, Werner PC, Pipp TL, Wilmot CB. Nutritional and metabolic response to acute spinal-cord injury. JPEN J Parenter Enteral Nutr. 1992 Jan-Feb;16(1):11-5. doi: 10.1177/014860719201600111. PMID 1738212
- [Background] Furuno K, Goodman MN, Goldberg AL. Role of different proteolytic systems in the degradation of muscle proteins during denervation atrophy. J Biol Chem. 1990 May 25;265(15):8550-7. PMID 2187867
- [Background] Cardus D, McTaggart WG. Body sodium and potassium in men with spinal cord injury. Arch Phys Med Rehabil. 1985 Mar;66(3):156-9. PMID 3977567
- [Background] Jacobs PL, Nash MS, Rusinowski JW. Circuit training provides cardiorespiratory and strength benefits in persons with paraplegia. Med Sci Sports Exerc. 2001 May;33(5):711-7. doi: 10.1097/00005768-200105000-00005. PMID 11323537
- [Background] Jacobs PL, Mahoney ET, Nash MS, Green BA. Circuit resistance training in persons with complete paraplegia. J Rehabil Res Dev. 2002 Jan-Feb;39(1):21-8. PMID 11926325
- See also: Center of Excellence in Functional Recovery in Chronic Spinal Cord Injury — http://www.sfvafre.org